CLINICAL TRIAL: NCT07277361
Title: Study of the Quality of Life of Patients With Fabry Disease Aged 65 and Over With and Without Specific Treatment
Acronym: FABRY65
Status: Recruiting | Type: Observational
Sponsor: Wladimir MAUHIN, Dr (Other)
Collaborators: University Hospital, Angers (Other Government); University Hospital, Bordeaux (Other); Centre Hospitalier Bretagne Atlantique (Other); Centre Hospitalier Universitaire de Caen (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Lille (Other); University Hospital, Limoges (Other); University Hospital, Marseille (Other); Nantes University Hospital (Other); Necker Hospital, 75015 Paris (Unknown); Rennes University Hospital (Other); University Hospital, Tours (Other); Hôpital Raymond Poincaré (Other); University Hospital, Rouen (Other); Hospital, Vannes (Unknown); University Hospital, Brest (Other); University Hospital, Grenoble (Other); University Hospital, Strasbourg (Other); Hospices Civils de Lyon (Other); Centre Hospitalier de la côte Basque (Other); University Hospital, Montpellier (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor-Investigator, Wladimir MAUHIN, Dr, Internist, Groupe Hospitalier Diaconesses Croix Saint-Simon
Organization: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Other Study IDs: GHDCSS_Non-RIPH-MI_3_2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Fabry Disease; Aged 65 Years or Older; Alpha Galactosidase A Deficiency; Galactosidase A Gene Mutation
Keywords: Fabry disease; Alpha galactosidase A deficiency
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants aged 65 or over with Fabry disease

SUMMARY:
Fabry disease is a rare genetic disorder affecting 1 in 10,000 individuals, leading to complications such as chronic pain, heart and kidney failure, and strokes, ultimately impacting life expectancy. People with this disease are increasingly being diagnosed later in life, around the age of 65, as the condition progresses slowly with irreversible organ damage. The effectiveness of treatments for Fabry disease remains controversial, but early initiation is recommended for long-term benefits. Despite the high cost and inconvenience of treatments, there is limited research on their efficacy in older people or on the quality of life for those aged 65 and over with Fabry disease. This study aims to assess the quality of life in this age group both with and without treatment over a period of 5 years to determine the benefits of treatment beyond the age of 65.

DETAILED DESCRIPTION:
Fabry disease is an X-linked genetic lysosomal disorder with an estimated prevalence of 1 in 10,000. It affects quality of life and life expectancy, through, among other things, chronic pain and the development of heart and kidney failure and stroke. An increasing number of people are being diagnosed at around the age of 65 or even later. Fabry disease develops slowly and progressively, causing irreversible organ damage. While the efficacy of Fabry disease treatments is debated, it is expected that they will be effective in the long term, provided therapy is initiated early.

Currently, there are no specific studies evaluating the efficacy of these treatments in people aged 65 and over. These treatments are very expensive (averaging €200k per individual treated per year) and sometimes cumbersome (involving twice-monthly infusions lasting several hours). There are also no studies on the quality of life of the people aged 65 and over with Fabry disease.

Furthermore, there is no clear evidence of any benefit from introducing or continuing treatment beyond the age of 65.

Our aim is to evaluate the quality of life of participants with Fabry disease aged 65 and over, both with and without treatment, at baseline and at 2 and 5 year intervals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 and over with a diagnosis of Fabry disease with, for men, a proven alpha-galactosidase A deficiency or an identified pathogenic GLA genetic variant, and for women, an identified pathogenic GLA variant.
* Minimum work-up available: ECG, 24h holterECG, cardiac ultrasound, creatinemia, proteinuria and/or microalbuminuria.
* Have received written and oral information about the protocol and have not expressed any opposition to participating in the study.
* Affiliated to a social security scheme or entitled to benefits (excluding AME).

Exclusion Criteria:

* Inability to understand the information provided,
* Under guardianship, curatorship or safeguard of justice,
* Under restraint or deprived of liberty by judicial or administrative decision.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People, men and women aged 65 and over, with a diagnosis of Fabry disease with for men, a proven alpha-galactosidase A deficiency or an identified pathogenic GLA genetic variant, and for women, an identified pathogenic GLA variant.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2029-10-14 (Estimated); Study Completion 2031-10-14 (Estimated)

PRIMARY OUTCOMES:
Evolution of quality of life assessed by the EQ-5D-5L score according to the existence or not of a specific treatment at 5 years in Fabry patients aged 65 and over. | 5 years
  People diagnosed with Fabry disease, will be evaluated for their quality of life, using a questionnaire based on the European Quality Of Life 5 Dimensions and 5 Lines (EQ-5D-5L) score, at baseline, 2 years and 5 years.
  The EQ-5D-5L score is an European quality of life scale. It is presented as follows: a first part with questions known as the 'EQ-5D descriptive system', supplemented by a visual analogue scale known as the 'EQ-5D VAS'.
  For the first part, the answers are given on 5-point scales (1: no problem; 2: slight problems; 3: moderate problems; 4: severe problems; 5: extreme problems or total incapacity).
  For the second part, it consists of a 20 cm line, graduated from 0 to 100, on which the participant must indicate how he or she rates his or her current state of health, 0 being the worst possible state and 100 the best.

SECONDARY OUTCOMES:
Identify the occurrence of a severe clinical or biological event since inclusion (cardiac rhythm disorder requiring the introduction of treatment or equipment, occurrence of a transient or permanent stroke, deterioration in creatinine clearance > 30%). | Year 2 and year 5
Identify the medical and social risk factors, whether related to the disease or not, associated with the lack of improvement in quality of life or the occurrence of an event (correlation and cluster studies) | Year 2, year 5
Evaluation of quality of life at baseline and 2 years. | Day 0 and year 2
  People diagnosed with Fabry disease, will be evaluated for their quality of life, using a questionnaire based on the European Quality Of Life 5 Dimensions and 5 Lines (EQ-5D-5L) score, at baseline and 2 years. The EQ-5D-5L score is an European quality of life scale. It is presented as follows: a first part with questions known as the 'EQ-5D descriptive system', supplemented by a visual analogue scale known as the 'EQ-5D VAS'.
  For the first part, the answers are given on 5-point scales (1: no problem; 2: slight problems; 3: moderate problems; 4: severe problems; 5: extreme problems or total incapacity).
  For the second part, it consists of a 20 cm line, graduated from 0 to 100, on which the participant must indicate how he or she rates his or her current state of health, 0 being the worst possible state and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Wladimir MAUHIN, Doctor, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided